CLINICAL TRIAL: NCT00687349
Title: Improving Patient Outcomes in End-of-Life Care Provided by Physicians and Nurses
Brief Title: Improving Clinician Communication Skills (ICCS)
Acronym: ICCS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, J. Randall Curtis, Professor of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 31466-G; R01NR009987 (NIH)
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Advanced Cancer; Chronic Obstructive Pulmonary Disease (COPD); Restrictive Lung Disease; Congestive Heart Failure; End Stage Liver Disease
Keywords: End-of-Life issues; Talking with your doctor; Coping with chronic illness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; End Stage Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Arm (Experimental): The training program will assign resident or NP student to a rotation. They will be receiving the educational intervention during 8 half-day sessions.
  Interventions: Behavioral: Training Program Intervention
- Control Arm (No Intervention): Resident or NP student is assigned to usual education.

INTERVENTIONS:
Behavioral: Training Program Intervention — Resident or NP Student receives the educational intervention during 8 half-day sessions.
  Arms: Intervention Arm

SUMMARY:
This research study is a randomized trial to evaluate a training program that is designed to improve the communication skills of clinicians. The training program focuses on care for patients with serious illnesses and their family members, and assesses effectiveness using patient and family outcomes. The long term goal of this research is to improve communication skills of doctors and nurses, thereby improving patient and family outcomes.

DETAILED DESCRIPTION:
Three decades of research on end-of-life care in the United States indicates that people who are dying often spend their final days with a significant burden of pain and other symptoms and receive care they would not choose. Patient-clinician communication about end-of-life care is an important focus for improving patient-centered end-of-life care for three reasons: 1) it is an integral component of clinician skill that affects all other aspects of end-of-life care; 2) physicians and nurses in practice do not demonstrate adequate skills for communicating about end-of-life care; and 3) current training in end-of-life communication is inadequate. Studies have shown that clinicians can improve their communication skills with experiential training, but no studies to date have shown that an intervention to improve clinician communication skill improves patient outcomes. Furthermore, despite widespread knowledge that end-of-life care is best delivered in an interdisciplinary context, most studies do not incorporate interdisciplinary training that includes physicians and nurses.

This is a randomized trial of a communication skills workshop for internal medicine residents and nurse practitioner (NP) students. A total of 373 residents and 128 NP students from two large training programs (UW and MUSC) will be randomized to either the intervention or usual education. The study's primary outcome measure will be the QOC scores on the "communication about end-of-life care" domain. The QOC will be assessed by patients, family members, and nurses before and after the intervention time period for all trainees. Secondary outcome measures are patient symptoms and patient-, family - and nurse-assessed QEOLC scores. Outcome measures will be collected for 5 patients and family members per trainee before the intervention period and 5 patients and family members per trainee after the intervention period. Process measures for both residents and NP students will include pre- and post-intervention assessment of knowledge, attitudes, and behavior regarding communication using standardized patient assessment as well as self-assessment and faculty assessment.

ELIGIBILITY:
Inclusion Criteria:

Physician:

* all internal medicine residents at either University of Washington (UW)or the Medical University of South Carolina
* who have a clinical rotation allowing implementation of the intervention.

NP Student:

* All NP Students at UW or MUSC
* in programs that train them to work with the following patient types:
* Adult patents with Cancer or other chronic, life-limiting illnesses
* Older Adults
* Adults Primary Care Patients

Patient:

One or more of the following diagnostic criteria:

* Advanced Cancer;
* Chronic obstructive pulmonary disease (COPD) with FEV1 values < 35% predicted and/or oxygen dependent;
* Restrictive lung disease with a TLC < 50% predicted;
* Congestive heart failure with an ejection fraction <30% or functional deficits matching New York Heart Association Class III or IV heart failure;
* End stage liver disease including Child's Class C cirrhosis, MELD score ≥ 18, a variceal bleed, refractory ascites, or spontaneous bacterial peritonitis (SBP);
* a Charlson Comorbidity Score point value ≥6;
* in-patients with a University HealthSystem Consortium (UHC) Risk of Mortality score of major or extreme;
* OR hospitalized patients ≥ 80 years.

Family:

* The ability to speak English well enough to be able to complete the study procedures
* AND no significant dementia or delirium that would limit the family member's ability to complete instruments.

Nurse-evaluators:

* are working in the hospital or clinic with the resident or NP student enrolled in the study.

Exclusion Criteria:

* less than 18 years,
* significant dementia, delirium, or psychosis;
* the inability to speak English well enough to be able to complete the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6086 (Actual)
Dates: Start 2007-04; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Patient and family ratings on the "End-of-Life domain" of the Quality of Communication Questionaire (QOC) | 4/1/2007-3/31/2012

SECONDARY OUTCOMES:
Patient symptoms of depression as assessed by the PHQ-8 (Memorial Symptom Assessment scale) | 4/01/2007-3/31/2012
Patient-, family-, and nurse-assessed ratings of the quality of end-of-life care provided by study clinicians using Quality of End-of-Life Care questionaire | 4/01/2007-3/31/2012

CONTACTS AND LOCATIONS:
Overall Officials: J. Randall Curtis, MD, MPH, Principal Investigator — University of Washington, Div. of Pulmonary and Critical Care Medicine
Locations (4):
- United States (4):
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Washington; Harborview Medical Center, Seattle, Washington
  - Veteran's Affairs Puget Sound HCS, Seattle, Washington
  - University of Washington; UW Medical Center, Seattle, Washington

REFERENCES:
- [Result] Curtis JR, Back AL, Ford DW, Downey L, Shannon SE, Doorenbos AZ, Kross EK, Reinke LF, Feemster LC, Edlund B, Arnold RW, O'Connor K, Engelberg RA. Effect of communication skills training for residents and nurse practitioners on quality of communication with patients with serious illness: a randomized trial. JAMA. 2013 Dec 4;310(21):2271-81. doi: 10.1001/jama.2013.282081. PMID 24302090
- [Derived] Ford DW, Downey L, Engelberg R, Back AL, Curtis JR. Association between Physician Trainee Self-Assessments in Discussing Religion and Spirituality and Their Patients' Reports. J Palliat Med. 2014 Apr;17(4):453-62. doi: 10.1089/jpm.2013.0388. Epub 2014 Mar 20. PMID 24649963